CLINICAL TRIAL: NCT07320014
Title: Inflammatory Profile in Patients Hospitalized for Heart Failure With Preserved or Mildly Reduced Ejection Fraction and Its Correlation With Bioimpedance Parameters and Other Biomarkers With Prognostic Value
Brief Title: Descriptive Study of Circulating Gene or Protein Inflammatory Biomarkers and Bioimpedance Parameters in a Population of Patients Hospitalized for Decompensated Heart Failure With Preserved or Mildly Reduced Cardiac Function
Acronym: BIOFEVIP
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Ana María Venegas Rodriguez, Cardiologist, M.D., Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: PIC011-25_FJD
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Inflammation Biomarkers; Heart Failure
Keywords: inflammatory profile; heart failure with preserved ejection fraction; heart failure with mildly reduced ejection fraction; bioimpedance
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected in EDTA tubes and immediately centrifuged and stored after extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Inflammatory biomarker sample collection — This is a prospective observational study in which a blood sample and a urine sample will be taken from all subjects in the first hours after admission. In addition, all subjects will be asked for specific consent for the isolation of plasma protein and nucleic acid (DNA/RNA). In addition, an echocardiogram and bioimpedance analysis will be performed in all patients included in the study.

SUMMARY:
The goal of this observational study is to determine whether changes in the inflammatory profile of heart failure patients can help identify those who may have a worse prognosis or who might benefit more from specific treatments. In addition, we aim to explore whether certain genes or gene mutations are related to a higher risk of future cardiovascular problems.

Heart failure continues to be a major cause of hospital admissions and death in our society. Because of this, it is very important for healthcare professionals to identify which patients are at higher risk of complications, so that we can provide the best possible treatment and follow-up. One method we use to help predict how the disease may evolve is the study of biomarkers, which are measurable biological substances that can help detect, monitor, or treat illnesses in a more personalized way.

In this study, the investigators will measure mainly inflammatory biomarkers that will be analyzed from a blood sample taken during hospital stay after being diagnosed with heart failure with preserved or mildly reduced ejection fraction. Any important health events that happen during the next six months after patients are discharged from hospital will also be recorded.

In addition, it is known that more than 2,000 diseases are known to be caused by changes in specific genes. In the case of cardiomyopathies-heart muscle diseases that can lead to heart failure-genetic causes vary depending on the type, and studies suggest that between 10% and 50% of cases may have a genetic origin. Identifying genetic markers linked to heart failure with preserved or mildly reduced ejection fraction may help improve prevention, treatment, and risk assessment, as some genetic changes may be associated with repeated cardiovascular events. By studying not only circulating biomarkers but also genetic factors, the investigators hope to better understand whether certain gene alterations may increase a person's tendency to experience additional heart-related events.

This is an observational study, which means that medical care and treatment will be exactly the same whether patients choose to participate or not. Participation involves allowing researchers to collect relevant information from medical records and agreeing to the collection of two or three small additional blood samples for research purposes. These samples will be used to measure the biomarkers and to analyze genes in the white blood cell fraction obtained from the same tubes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at recruitment.
* Signed informed consent.
* Hospitalization due to decompensated heart failure, based on Framingham criteria and elevated natriuretic peptides (N-terminal of the prohormone brain natriuretic peptide (NT-proBNP) ≥450 pg/ml, or ≥900 pg/ml for patients with atrial fibrillation or flutter).
* Left ventricular ejection fraction(LVEF) ≥40% and evidence of structural heart disease based on the presence of at least one of the following imaging criteria:

  * Left atrial dilation: LA diameter ≥3.8 cm, or area ≥20 cm², or LA volume ≥55 ml, or indexed LA volume ≥29 ml/m².
  * Left ventricular hypertrophy, defined as septal or posterior wall thickness ≥1.1 cm.
  * Evidence of increased filling pressures, measured by septal or lateral E/e' ratio >15 or >12, respectively.

Exclusion Criteria:

* Hemodynamic instability at the time of inclusion.
* Heart failure secondary to acute myocardial infarction (AMI).
* Pregnant or breastfeeding women.
* Comorbidities that could influence the clinical course:

  * COPD requiring long-term home oxygen therapy, oral corticosteroids, hospitalization due to exacerbation, or primary pulmonary arterial hypertension.
  * Chronic treatment with immunosuppressants, corticosteroids, or IL-1 antagonists within the 6 months prior to inclusion.
  * Confirmed active infection or patients currently receiving antibiotic treatment.
  * Acute or chronic liver disease.
  * Chronic kidney disease with eGFR <15 ml/min/1.73 m² or need for dialysis during hospitalization.
  * Hematological disorders, such as blood dyscrasias or hemoglobin <9 g/dl on admission.
  * Active oncological disease, except treated basal cell carcinoma or low-risk prostate cancer.
  * Patients with limb amputation or carriers of pacemakers or defibrillators (due to possible errors in BIA measurements).
  * Any disease associated with a life expectancy of less than one year, or patients expected to have difficulty adhering to the study protocol
* Patients actively participating in other clinical trials involving investigational drugs at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized for HF at the FundaciJiménez Díaz University Hospital (Madrid), with preserved or slightly reduced LV ejection fraction (LVEF ≥40%), with evidence of structural heart disease (left atrial dilation or left ventricular hypertrophy) and elevated natriuretic peptides.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Description of circulating inflammatory gene or protein biomarkers and other biomarkers with prognostic value in a population of patients hospitalized for acute HF. | At enrollment
  Biomarkers with prognostic value in heart failure such as troponins, natriuretic peptides or CA-125, biomarkers of mineral metabolism and inflammatory or profibrotic biomarkers including C- reactive protein, tumoral necrosis factor-α, interleukins, galectin-3, MCP-1, pentraxin-3 or myeloperoxidase, will be measured at admission in a population of patients hospitalized for decompensated heart failure with preserved or mildly reduced left ventricular ejection fraction.
Description of parameters obtained by bioimpedance analysis (BIA) in a population of patients hospitalized for decompensated HF with preserved or mildly reduced ejection fraction. | At enrollment
  Description of parameters obtained by bioimpedance analysis, including the assessment of body composition, hydration status and nutritional status in a population of patients hospitalized for decompensated HF with preserved or mildly reduced ejection fraction.

SECONDARY OUTCOMES:
Incidence of major cardiovascular events in a population of patients hospitalized for decompensated HF with preserved or mildly reduced LV ejection fraction and its correlation with the inflammatory status. | From inclusion to 6 months after discharge
  Description of the incidence of all-cause mortality, cardiovascular mortality, heart failure hospitalization or Emergency-Department visit requiring intravenous diuretics in the first 6 months after discharge in a population of patients hospitalized for decompensated HF with preserved or mildly reduced LV ejection fraction and its correlation with the inflammatory status.
Prognostic correlation of inflammatory biomarkers with the parameters obtained by bioimpedance analysis. | At enrollment
  To evaluate the prognostic correlation of inflammatory biomarkers measured in patients hospitalized for decompensated HF with preserved or mildly reduced LV ejection fraction with the parameters obtained by bioimpedance analysis performed at the time of inclusion, including both hydration and nutritional status.
Correlation of inflammatory biomarkers with other circulating biomarkers with prognostic value in HF. | At enrollment
  To study the correlation of the inflammatory profile alterations with other biomarkers with prognostic value in HF such as natriuretic peptides and fibrosis or mineral metabolism biomarkers.
Correlation of inflammatory biomarkers with echocardiographic data with prognostic value | At enrollment
  To examine the correlation of inflammatory biomarkers with echocardiographic study at enrollment, including left ventricular ejection fraction (LVEF), valvular heart disease, left ventricular end-diastolic diameter, myocardial wall thickness, left ventricular mass, parameters of left atrial dilation, right ventricular size and function, and parameters related to diastolic function.
Identification of different patient subgroups according to prognosis based on the inflammatory study. | From inclusion to 6 months after discharge
  To describe patient subgroups with different prognosis according to the etiology of heart failure or its associated comorbiditiesbased on the alterations identified in the inflammatory study.

IPD SHARING:
Plan to Share IPD: No